CLINICAL TRIAL: NCT04449848
Title: The Effect of Patient's Position After Intra-tympanic Injection on the Amount of Fluid in the Middle Ear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0182-20
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Sudden Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sitting after intra tympanic injection (Experimental): Patients with Sudden hearing loss sitting after intra tympanic injection of steroids
  Interventions: Other: Sitting after intra tympanic injection

INTERVENTIONS:
Other: Sitting after intra tympanic injection — Sitting after intra tympanic injection

SUMMARY:
During the regular protocol of Intra-tympanic injections of Dexamethasone to the middle ear due to Sudden Sensorineural Hearing Loss, the patients will be sitted once after the injection instead of lying down. They will be then asked to rate their taste as a reference to the amount of fluid leaking to the throat through the eustachian tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Sudden Sensorineural Hearing Loss, treated using intra-tympanic injection of steroids to the middle ear

Exclusion Criteria:

* Patients with abnormal sense of taste
* Middle or inner ear anomaly
* Eustachian tube dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Bitter taste | 30 minutes
  Bitter taste described by the patients using a questionnaire with a scale of 0 to 5

IPD SHARING:
Plan to Share IPD: No